CLINICAL TRIAL: NCT07041879
Title: Piezotome Atraumatic Tooth Extraction And Immediate Implant Placement In Maxillary Anterior Region: Randomized Clinical Trial
Brief Title: Piezotome Atraumatic Tooth Extraction And Immediate Implant Placement In Maxillary Anterior Region
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATE-17-5-25
Record Dates: First submitted 2025-05-17; First posted 2025-06-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-05

CONDITIONS: Piezotome; Implant-supported Single Crowns
Keywords: tooth extraction; immediate implant; bone healing; piezotome

STUDY DESIGN:
Intervention Model Description: Patients with maxillary anterior teeth will be atraumatically extracted with piezotome extraction kit, and subsequently immediate implant placement
Who Masked: Participant
Masking Description: Sequentially numbered, opaque, sealed envelopes (SNOSE) allocation concealment method will be utilized. Each participant included in the study will be given a serial number that will be used in the allocation. These numbers will be written in identical sheets of paper with the group to which each participant is allocated and placed inside opaque envelopes carrying the respective names of participants. A trial independent personnel will be assigned the role of keeping the envelopes and unfolding them only at the time of the operation, so that the participant is allocated to a group which is concealed from the operator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atraumatic extraction with piezotome and subsequently immediate implant placement (Active Comparator): Patients with maxillary anterior teeth will be atraumatically extracted with piezotome extraction, and subsequently immediate implant placement
  Interventions: Procedure: maxillary anterior teeth atraumatically extracted with piezotome extraction kit, and subsequent immediate implant placement
- Atraumatic extraction with periotome and subsequently immediate implant placement (Experimental): Patients with maxillary anterior teeth will be atraumatically extracted with periotome, and subsequently immediate implant placement
  Interventions: Procedure: maxillary anterior teeth atraumatically extracted with periotome, and subsequent immediate implant placment

INTERVENTIONS:
Procedure: maxillary anterior teeth atraumatically extracted with piezotome extraction kit, and subsequent immediate implant placement — piezotome extraction kit,
  Arms: Atraumatic extraction with piezotome and subsequently immediate implant placement
Procedure: maxillary anterior teeth atraumatically extracted with periotome, and subsequent immediate implant placment — periotome
  Arms: Atraumatic extraction with periotome and subsequently immediate implant placement

SUMMARY:
Tooth extraction is critical for dental treatment complications followed by immediate implant placement to restore the extracted tooth . The use of devices or instruments such as piezotome and periotome as aids in atraumatic surgical proceduresو conserving both bone and soft tissue, allowing extraction without unnecessary socket expansion. Immediate implant placement into fresh extraction sockets offers some esthetic and functional advantages.

the Aim of this study is to compare and evaluate the effectiveness of the piezotome and periotome as aids for atraumatic extraction in immediate implant placement in maxillary anterior teeth.

DETAILED DESCRIPTION:
30 patients with non-restorable maxillary anterior teeth will be included. Teeth will be extracted using an atraumatic tooth extraction using piezotome and periotome as aids in atraumatic surgical procedures. After that an immediate implant will be placed into the fresh extraction socket . patients will be recalled for follow-up 3months after implant placement to evaluate pain by VAS and evaluate bone healing using CBCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both gender with a non-restorable maxillary anterior tooth in the aesthetic zone indicated for extraction and subsequent immediate implant placement. Including those with:

   1. Severely carious tooth that it cannot be restored.
   2. Pulpal necrosis or irreversible pulpitis that is not amenable to endodontics.
   3. Periodontally involved Tooth with grade 2 mobility or above.
   4. Tooth with root caries that can't be restored.
2. Patients with extraction socket Type I, according to Elian's classification

Exclusion Criteria:

1. Patients with extraction socket Type II or III, with defect in the buccal plate
2. Patients with deciduous teeth.
3. Heavy smokers.
4. Medically compromised patients with conditions that would impede implant osteointegration and healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic assessment of the management of the crestal bone width and changes in labial bone thickness. | 5 months
  A postoperative CBCT will be taken within 24 hours of implant placement followed by a 6-months scan, and values will be compared with the preoperative record. The assessment will be conducted using the tools on the "On Demand 3D App." Software*. The following criteria will be assessed:

SECONDARY OUTCOMES:
Clinical Wound Healing | 21 days
  All patients will be recalled for a clinical follow-up period at 7, 14, and 21 days postoperative for the assessment of Wound healing using the Pink Esthetic Score (PES)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study